CLINICAL TRIAL: NCT03589079
Title: Delineation of Novel Monogenic Disorders in the United Arab Emirates
Brief Title: Delineation of Novel Monogenic Disorders in the United Arab Emirates Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IREC038
Record Dates: First submitted 2018-07-02; First posted 2018-07-17 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Mendelian Disorders; Genetic Disorder; Novel Mutation; Hereditary Disorder; De Novo Mutation; Inherited Disease; Single-Gene Defects
Keywords: Monogenic Disorder; Mendelian Disease; Single Gene Disorder; Next Generation Sequencing; Genetic testing
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA will be extracted from collected blood samples for genetic analysis

GROUPS / COHORTS (1):
- Monogenic Disorder: Participants exhibiting clinical phenotypes suggestive of an underlying novel monogenic disorder, with/without the presence of familial recurrence of the phenotype and/or parental consanguinity will be included. Sanger and/or Next generation Sequencing (NGS) - Panel/WES/WGS approaches will be used to facilitate identification of de novo/inherited variants in the child/proband.
  Interventions: Genetic: Sanger and/or Next Generation Sequencing (NGS)

INTERVENTIONS:
Genetic: Sanger and/or Next Generation Sequencing (NGS) — NGS panel, whole exome / genome sequencing (WES/WGS)

SUMMARY:
The study aims to identify novel monogenic phenotypes from specific pedigrees and discover the underlying causal genetic variant using genetic sequencing (Sanger and/or Next Generation Sequencing - Panel/WES/WGS) methodologies in families across the United Arab Emirates (UAE).

DETAILED DESCRIPTION:
Monogenic disorders result from a single defective gene and are inherited according to Mendel's Laws (Mendelian disorders). Such gene defects arise from a mutation that can either be inherited or occur spontaneously; both may occur in the absence of a previous family history. Inherited mutations can be dominant or recessive, and autosomal or sex-linked. According to WHO, although individually rare, collectively monogenic disorders affect millions of people worldwide. Currently, over 10,000 human diseases are estimated to be monogenic. Until recently the identification of the genetic causes, especially of extremely rare phenotypes, has not been possible or cost effective due to the scientific challenges of identifying causative mutations through linkage analysis. The advent of cost effective next generation sequencing now facilitates the identification of all rare variants across the whole genome, in turn allowing mutation identification in small families and, if de novo, even in single cases.

The clinical application of single gene sequencing potentially provides tangible benefits to patients, informing diagnosis and prognosis, and may guide treatment choice. Next generation sequencing (NGS) panels sequence multiple genes in parallel and are now entering the clinical domain. NGS provides significant advantages over single gene sequencing for conditions which are genetically heterogeneous, such as the epilepsies. However, as more genes are included in an NGS panel, the possibility of incidental findings rises significantly, with associated challenges in result interpretation. Since many conditions are phenotypically as well as genetically heterogeneous, acquisition of detailed phenotypic information is essential for meaningful interpretation of NGS results.

Monogenic (Mendelian) disorders have historically provided the clearest means of elucidating human gene function. The linkage of a rare DNA variant to altered protein function or dose to discrete phenotype has important implications for fundamental biology, monogenic disease pathogenesis, complex traits, diagnostics and therapy. By representing the most readily interpretable component of human genetics in defining a clear, high-penetrance phenotype arising from alteration in function of a single gene, study of monogenic disorders can identify the genetic basis for novel or existing phenotypes and provide insights into non-redundant biological pathways that may inform therapeutic targeting for both the specific rare variant and common diseases. Accordingly the primary purpose of this programme is to identify novel monogenic phenotypes and discover underlying causal genetic variants by genetic sequencing in families across the UAE.

ELIGIBILITY:
Inclusion Criteria:

* Specific phenotype - Phenotypes of interest suggestive of an underlying novel genetic disorder:

  1. Unusual presentations of common disorders, e.g. with clearly defined syndromic/dysmorphic features*.
  2. Extreme phenotypic presentations.
  3. Entirely novel, previously undefined phenotypes.
* Family history/pedigree - Phenotype suspected to be due to a single genetic mutation (de novo or inherited) based, where available, on any of:

  1. Presence of syndromic/dysmorphic features.
  2. Family history of similar presentations in other relative(s).
  3. Pattern of inheritance.
  4. Parental consanguinity.
* Clinical interpretation - Where available (i.e. not mandatory but will increase confidence in suitability), the presence of clinical and/or investigation results consistent with a novel inherited/monogenic disorder:

  1. Exclusion of non-genetic acquired causes - e.g. those with a clear history of likely environmental cause.
  2. Genotype negative for known genes underlying the disorder/phenotype.
* Consent - Participant (or parent/legal guardian if aged under 18 years) willing and able to give informed consent for participation in the study as the proband (male/female), parent in a trio or extended family member.

Exclusion Criteria:

* Participant or their legal guardian/legal representative is unwilling or unable to give informed consent. In cases where a potential child participant has capacity to assent but refuses to participate, the will of the child will be respected.
* Participant who has already undergone genotyping/panel/laboratory testing (e.g. for known inborn errors of metabolism) and has a defined/diagnosed genetic condition.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be exhibiting clinical phenotypes suggestive of an underlying novel monogenic disorder, with/without the presence of familial recurrence of the phenotype and/or parental consanguinity.
  Pedigrees of particular interest (in order of preference) will include:
  * Consanguineous families, ideally where one or more family member is affected
  * De novo based - i.e. trios of proband and both parents, where only the proband exhibits the phenotype
  * Autosomal recessive
  * Autosomal dominant, albeit with a large kindred (e.g. ideally 6-8 affected members across 2-3 generations)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Novel phenotype and gene discovery | through study completion, an average of 2 year
  Identification and characterisation of novel monogenic phenotypes from specific pedigrees.
  Unbiased identification of novel, rare disease-causing genes through application of genetic sequencing methodologies to new or established phenotypes.

SECONDARY OUTCOMES:
Generate new biological insights | through study completion, an average of 2 year
  Obtain insights into the pathological mechanisms (known or new downstream disease pathways) underlying monogenic disease and more broadly to common/complex diseases, in addition to fundamental insights concerning physiological gene function.
Modifier genes of monogenic disorders | through study completion, an average of 2 year
  Identify modifier genes of monogenic disorders - to aid understanding of phenotypic heterogeneity of Mendelian disorders.
Potential new therapeutic targets | through study completion, an average of 2 year
  Identify potential new therapeutic targets - leverage these insights to identify robust, genetically-defined potential molecular and cellular drug targets (related to the primary gene and/or modifier genes) for the treatment of rare (orphan) and/or common disease.
Gene function and target validation | through study completion, an average of 2 year
  Where feasible, determine the functional impact of identified pathogenic variants and validate disease mechanism-based targets through the use of pre-clinical (in vitro/in vivo) and/or early human experimental studies.

CONTACTS AND LOCATIONS:
Overall Officials: Maha Barakat, PhD FRCP, Principal Investigator — Imperial College London Diabetes Centre; Houman Ashrafian, DPhil FRCP, Principal Investigator — University of Oxford
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] 1- Chial H. Rare Genetic Disorders: Learning About Genetic Disease Through Gene Mapping, SNPs, and Microarray Data. Nature Education 2008;1(1):192.
- [Background] 2- Genes and human disease. World Heath Organization 2017. Retrieved from http://www.who.int/genomics/public/geneticdiseases/en/index2.html
- [Background] Ku CS, Cooper DN, Patrinos GP. The Rise and Rise of Exome Sequencing. Public Health Genomics. 2016;19(6):315-324. doi: 10.1159/000450991. Epub 2016 Nov 30. PMID 27898412
- [Background] Mefford HC. Clinical Genetic Testing in Epilepsy. Epilepsy Curr. 2015 Jul-Aug;15(4):197-201. doi: 10.5698/1535-7511-15.4.197. PMID 26316867
- [Background] de Ligt J, Willemsen MH, van Bon BW, Kleefstra T, Yntema HG, Kroes T, Vulto-van Silfhout AT, Koolen DA, de Vries P, Gilissen C, del Rosario M, Hoischen A, Scheffer H, de Vries BB, Brunner HG, Veltman JA, Vissers LE. Diagnostic exome sequencing in persons with severe intellectual disability. N Engl J Med. 2012 Nov 15;367(20):1921-9. doi: 10.1056/NEJMoa1206524. Epub 2012 Oct 3. PMID 23033978
- [Background] Della Mina E, Ciccone R, Brustia F, Bayindir B, Limongelli I, Vetro A, Iascone M, Pezzoli L, Bellazzi R, Perotti G, De Giorgis V, Lunghi S, Coppola G, Orcesi S, Merli P, Savasta S, Veggiotti P, Zuffardi O. Improving molecular diagnosis in epilepsy by a dedicated high-throughput sequencing platform. Eur J Hum Genet. 2015 Mar;23(3):354-62. doi: 10.1038/ejhg.2014.92. Epub 2014 May 21. PMID 24848745